## **Clinical Trial Protocol**

Patient-Customized Bioprinting Technology for Practical Regeneration of the Respiratory Tract (Trachea)

Protocol No. : 3D Bioprinting Trachea

Protocol Version : 2.3

Development date : 2023-05-26

## CLINICAL TRIAL PROTOCOL: CLINICAL RESEARCH PLAN OVERVIEW

| Professor Bae Ja-sung, Seoul St. Mary's Hospital | |
|---|---|
| Patient-Customized Bioprinting Technology for Practical 기톨릭대학교 서울성모병원 | |
| Regeneration of the Respiratory Tract (Trachea) | |
| Study Title | Patient-Customized Bioprinting Technology for Practical |
| | Regeneration of the Respiratory Tract (Trachea) |
| Principal | Professor Bae Ja-sung, Catholic University of Korea, Seoul St. Mary's Hospital |
| Investigator | |
| Clinical Research | Catholic University of Korea, Seoul St. Mary's Hospital |
| Institution | |
| Reference | Bae Ja-sung, et al. Rational Tissue Engineering Strategy for Extensive |
| | Circumferential Tracheal Reconstruction Using Three-Dimensional (3D) |
| | Printing. Biomaterials. 2018;185:276-283. |
| Period | 72 months from IRB approval <b>Stage</b> Cell therapy phase for |
| | date academic purposes |
| Objective | This clinical study aims to assess the effectiveness and safety of transplanting |
| | 3D patient-specific bioprinted tracheal organs using biopolymers, hydrogels, |
| | and tissue regeneration cells for respiratory tract regeneration. |
| Methods | Participants with thyroid or airway diseases necessitating partial or segmental |
| | resection will be enrolled after providing written consent. Screening tests will |
| | determine eligibility. The 3D bioprinted trachea, incorporating stem cells from |
| | the nasal cavity and nasal septum cartilage, will be transplanted. Evaluation |
| | includes endoscopy, bronchoscopy, CT, and lab tests. Neck fixing splints will |
| | stabilize transplanted areas post-surgery. Thyroid cancer patients will have |
| | extended follow-up with specific tests. |
| Number of | 1 |
| Participants | |
| Target Disease | Congenital tracheal softening, traumatic tracheal stenosis, tracheal defects |
| | post-thyroid cancer surgery, requiring partial or segmental resection |
| Selection/Exclusio | Selection Criteria: |
| n Criteria | Adults aged 19-75 |
| | Patients meeting criteria for thyroid or airway disease requiring resection |
| | Patients with thyroid cancer invading the trachea, requiring resection with |
| | expected organ dysfunction post-surgery |
| | <ul> <li>Patients with organ defects around cartilage (&gt;30%), suitable for 3D</li> </ul> |
| | bioprinting |
| | Female participants using contraception during the study |
| | Participants providing informed consent |

## **Protocol No. 3D Bioprinting Trachea**

| | Exclusion Criteria: |
|---|---|
| | Pregnant or lactating women |
| | Prior thyroid or airway peripheral surgery |
| | Inflammation of thyroid or surrounding tissues |
| | Systemic inflammatory disease |
| | High risk due to liver, kidney, or heart disease |
| | Sepsis or hemorrhagic predisposition |
| | Prior radiotherapy to head/neck |
| | Recent use of other research medications/devices |
| | History of cell therapy |
| | Malignant tumors other than thyroid cancer |
| | Other deemed inappropriate for the study |
| Product | 3D cell-printed trachea using patient-specific cells (hNTSCs, hNCs) and |
| Description | hydrogels |
| | Patient-specific single-product bioprinted trachea |
| | No artificial genetic manipulation |
| Validity | Primary Variables: |
| Assessment | • Endoscopic findings after 1, 2, 4, and 24 weeks |
| | Airway intraluminal clearance rate |
| | Degree of granuloma and bark formation |
| | Inflammation and other findings |
| | Secondary outcome |
| | CT-based airway condition comparison |
| | Postoperative inflammatory levels (WBC, WBC Diff, CRP, ESR) |
| | Bronchoscopy findings (wall stability, tracheal opening, mucosal formation, |
| | inflammation/granulation) |
| Safety | Abnormal management with signs FCC lab tasts about a law and |
| Assessment | Abnormal responses, vital signs, ECG, lab tests, physical exam |